CLINICAL TRIAL: NCT06141174
Title: Predictors of Outcome in Patients With Pleural Infection at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amany Eldawwy Hashem, resident at chest diseases and tuberculosis, Sohag University
Other Study IDs: Soh-med-23-10-08ms
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pleural Infection
MeSH Terms: interventions — Mortality; Length of Stay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: disease outcome ( mortality and length of stay ) — insertion of intercostal tube to drain pleural collection

SUMMARY:
pleural infection remains a common medical problem with significant mortality and morbidity despite a better undrstanding of the aetiology , pathophysiology and recent advances in management approaches .

the cornerstones of the managment op pleural infection include early identification of cases and accurate diagnosis . suitable antibiotic therapy , nutrition managment , efficient drainage of infected collection via chest tube with or without adjunctive therapies including intrapleural agents and ultimately surgical managment .

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years old with pleural infection

Exclusion Criteria:

* hemothorax
* chest trauma within 3 month
* underwent thoracic surgery within 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients more than 18 years old with pleural infection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
lenght of hospital stay | 1 month
  lenght of hospital stay since admission up to improvement

SECONDARY OUTCOMES:
mortality rate | up to 30 days , 3 months
  mortality rate related to pleural infection

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gould J. Pleural infection: a case where clinical improvement was misleading. BMJ Case Rep. 2013 Apr 18;2013:bcr2013008700. doi: 10.1136/bcr-2013-008700. PMID 23605824
- [Background] Rahman NM, Maskell NA, West A, Teoh R, Arnold A, Mackinlay C, Peckham D, Davies CW, Ali N, Kinnear W, Bentley A, Kahan BC, Wrightson JM, Davies HE, Hooper CE, Lee YC, Hedley EL, Crosthwaite N, Choo L, Helm EJ, Gleeson FV, Nunn AJ, Davies RJ. Intrapleural use of tissue plasminogen activator and DNase in pleural infection. N Engl J Med. 2011 Aug 11;365(6):518-26. doi: 10.1056/NEJMoa1012740. PMID 21830966
- [Background] Davies CW, Gleeson FV, Davies RJ; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of pleural infection. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii18-28. doi: 10.1136/thorax.58.suppl_2.ii18. No abstract available. PMID 12728147
- [Background] Davies HE, Davies RJ, Davies CW; BTS Pleural Disease Guideline Group. Management of pleural infection in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii41-53. doi: 10.1136/thx.2010.137000. No abstract available. PMID 20696693